CLINICAL TRIAL: NCT02806336
Title: Multimodel Exercise and Weight Loss in Older Obese Veterans With Dysmobility
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E1813-R; 1I01RX001813-01A1 (NIH)
Record Dates: First submitted 2016-06-02; First posted 2016-06-20 (Estimated); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Dysmobility
Keywords: exercise training; assistive device; weight loss; function; mobility
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Two group randomized control trial (RCT)
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded to group, statistical analyses blinded to group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi Modal Balance Training & Weight Loss (Experimental): Supervised exercise 3 times per week for about 1 hour. The classes will consist of a group balance class (about 30 minutes), a supervised obstacle course (about 10 minutes), and lower body and core body strength exercises (about 20 minutes). Weekly nutrition sessions for individual dietary recommendations designed to produce about a 10% weight loss over the first six months of the study.
  Interventions: Behavioral: Multi Modal Balance Training (MMBI); Behavioral: Weight Loss (WL)
- Multi Modal Balance Training Only (Active Comparator): Supervised exercise 3 times per week for about 1 hour. The classes will consist of a group balance class (about 30 minutes), a supervised obstacle course (about 10 minutes), and lower body and core body strength exercises (about 20 minutes).
  Interventions: Behavioral: Multi Modal Balance Training (MMBI)

INTERVENTIONS:
Behavioral: Multi Modal Balance Training (MMBI) — Group balance class, obstacle course, strengthening exercises
  Other Names: MMBI
Behavioral: Weight Loss (WL) — Nutritional counseling to achieve 500 kcal standard hypocaloric diet
  Other Names: WL
  Arms: Multi Modal Balance Training & Weight Loss

SUMMARY:
Obesity is a major risk factor for mobility problems in older adults and many older adults use a walking aid to help with their mobility. The use of a walking aid changes normal walking patterns and makes walking harder, leading people to have more functional problems. The purpose of this study is to test the effects of 12 months of a multi-modal balance intervention (MMBI) with supervised weight loss compared to MMBI only on fitness, functional performance, balance, and economy of gait. Participants will be one of 120 participants in the VA Maryland Health Care System (VAMHCS). Participation in this study is voluntary. The research will be conducted at the VAMHCS. The entire study will take approximately 4 years to complete. Subjects' participation in the study will last 24 months.

DETAILED DESCRIPTION:
Note: Study has been completed, enrollment and study interventions were severely impacted by coronavirus disease 2019 (COVID)

Older obese adults suffer disproportionately from walking mobility limitations. Sedentary, obese older adults are at an increased risk for having or developing difficulties with mobility. These individuals are often excluded from studies due to their advanced mobility limitations. A number of studies have compared the effects of weight loss alone, exercise alone, or weight loss in combination with exercise on functional performance in older adults, but none of the studies have specifically targeted subjects who use walking assistive devices. The purpose of this study is to test the effects of a 12 month multi-modal exercise rehabilitation intervention with a nutrition program versus a nutrition program only on fitness, functional performance, mobility, and muscle mass. The results of this study will lead to new and more effective interventions that could reduce disability, fall risk, injury-related hospitalization and death in older Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 60
* Body Mass Index (BMI) >= 30 kg/m2
* Dysmobility as define by 1 or more of the following: Use of or prescribed an assistive walking device, measured gait speed < 1.0 m/s, Four Square Step Test >/= 12 secs OR inability to complete the Four Square Step Test, and/or self-reported difficulty walking 1 km.
* Community dwelling

Exclusion Criteria:

* Unable to walk >0.2 mph on a treadmill for 2 minutes
* Poorly controlled hypertension >180 systolic or >100 diastolic
* Episodes of acute coronary syndrome, coronary revascularization, or major cardiac/vascular procedures within the prior 6 months
* New York Heart Association Class 3 or 4 heart failure
* Symptomatic angina at rest or during exercise
* Syncope within the past 12 months without known cause or resolution
* Chronic lung disease required oxygen dependency
* Severe spinal stenosis limiting ambulation
* Known dementia
* Mini Mental State Exam score <24
* Transtibial or above the knee amputation
* Currently enrolled and active in a supervised exercise program or Weight Management Program for Veterans (MOVE)
* Poorly controlled diabetes as defined by HbA1C >10% or frequent hypoglycemic episodes
* Currently undergoing chemotherapy and/or radiation therapy for cancer treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie I Katzel, MD PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were excluded from the study before assignment to groups due to the corona virus 19 (COVID-19) pandemic and associated research activity shut down.
Groups:
- Multi Modal Balance Training & Weight Loss: Supervised exercise 3 times per week for about 1 hour. The classes will consist of a group balance class (about 30 minutes), a supervised obstacle course (about 10 minutes), and lower body and core body strength exercises (about 20 minutes). Weekly nutrition sessions for individual dietary recommendations designed to produce about a 10% weight loss over the first six months of the study.
  Multi Modal Balance Training: Group balance class, obstacle course, strengthening exercises
  Weight Loss: Nutritional counseling to achieve 500 kcal standard hypocaloric diet
- Multi Modal Balance Training Only: Supervised exercise 3 times per week for about 1 hour. The classes will consist of a group balance class (about 30 minutes), a supervised obstacle course (about 10 minutes), and lower body and core body strength exercises (about 20 minutes).
  Multi Modal Balance Training: Group balance class, obstacle course, strengthening exercises
Period: Overall Study
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
Started | 9 | 11
Completed | 3 | 2
Not Completed | 6 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4
Not completed — COVID-19 research shut down | 3 | 4
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.44 (8.50) | 71.73 (5.37) | 71.15 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 11 | 20
Body Mass Index (BMI) (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 37.72 (4.84) | 36.65 (5.02) | 37.18 (4.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in 6 Minute Walk Distance
Description: Distance walked during the 6 minute walking test
Time Frame: 6 months
Population: There may have been certain circumstances in which the Principal Investigator or clinical investigative team chose not to perform some of the research procedures or there may have been unforeseen problems with data collection.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
Number analyzed (Participants) | 9 | 9
feet | 1137 (328) | 1195 (425)
Statistical Analysis 1: Comparison: Multi Modal Balance Training & Weight Loss vs Multi Modal Balance Training Only; change in combined groups; Test type: Superiority; p = 0.03, t-test, 2 sided

2. Secondary Outcome: Change in 6 Minute Walk With Oxygen Uptake (VO2) Measurement
Description: 6 minute walk with submaximal assessment of oxygen uptake as a measure of fitness.
Time Frame: 6 months
Population: There were certain circumstances in which the Principal Investigator or clinical investigative team chose not to perform some of the research procedures.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
Number analyzed (Participants) | 9 | 9
ml/kg/min | 13.46 (4.04) | 15.01 (3.64)
Statistical Analysis 1: Comparison: Multi Modal Balance Training & Weight Loss vs Multi Modal Balance Training Only; Test type: Superiority; p = 0.34, t-test, 2 sided

3. Secondary Outcome: Change in Lean Mass as Assessed by Dual Energy X Ray Absorptiometry (DXA) Scan
Description: The DXA scan provides information about the body composition including total body fat, and lean muscle mass
Time Frame: baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
Number analyzed (Participants) | 7 | 6
grams
  Baseline | 64185 (15175.8) | 66642.5 (4653.3)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 63251 (14811.1) | 69376.5 (4599.7)
Statistical Analysis 1: Comparison: Multi Modal Balance Training & Weight Loss vs Multi Modal Balance Training Only; Test type: Superiority; p = 0.78, t-test, 2 sided

4. Secondary Outcome: Change in Gait Biomechanics
Description: Gait biomechanics as assessed by walking mechanics on the gait rite mat. Scale range 0 - 24 with higher scores indicating better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
Number analyzed (Participants) | 9 | 9
score on a scale | 16.8 (6) | 20.3 (7)
Statistical Analysis 1: Comparison: Multi Modal Balance Training & Weight Loss; Test type: Superiority; p = 0.03, t-test, 2 sided — change in functional gait analysis (FGA) in combined groups compared to baseline

5. Secondary Outcome: Change in Short Physical Performance Battery
Description: overall short physical performance battery score. Scale range 0 - 12 with higher scores indicating better possible function.
Time Frame: baseline, 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
Number analyzed (Participants) | 7 | 7
units on a scale
  Baseline | 9 (2) | 9 (3)
  3 months: number analyzed (Participants) | 7 | 5
  3 months | 10 (2) | 11 (2)
Statistical Analysis 1: Comparison: Multi Modal Balance Training & Weight Loss vs Multi Modal Balance Training Only; Test type: Superiority; p = 0.14, t-test, 2 sided

6. Secondary Outcome: Change in Four Square Step Test
Description: Dynamic test of balance involving change in stepping direction.
Time Frame: baseline, 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
Number analyzed (Participants) | 7 | 7
seconds
  Baseline | 12.58 (3.06) | 17.68 (6.40)
  3 months: number analyzed (Participants) | 7 | 5
  3 months | 10.67 (1.63) | 11.69 (4.14)
Statistical Analysis 1: Comparison: Multi Modal Balance Training & Weight Loss vs Multi Modal Balance Training Only; Test type: Superiority; p = .17, t-test, 2 sided
Statistical Analysis 2: Comparison: Multi Modal Balance Training & Weight Loss vs Multi Modal Balance Training Only; Test type: Superiority; p = 0.14, t-test, 2 sided

7. Secondary Outcome: Change in 8 Foot up and go
Description: Time to get up from a chair and walk around a cone 8 feet away and sit back down, representing agility.
Time Frame: baseline, 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
Number analyzed (Participants) | 7 | 7
seconds
  Baseline | 9.00 (2.61) | 10.24 (3.12)
  3 months: number analyzed (Participants) | 7 | 5
  3 months | 9.78 (2.82) | 8.33 (2.34)
Statistical Analysis 1: Comparison: Multi Modal Balance Training & Weight Loss vs Multi Modal Balance Training Only; Test type: Superiority; p = 0.23, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: The definitions of adverse events and serious adverse events does not differ from the clinical trials definitions.
Arm/Group | Multi Modal Balance Training & Weight Loss | Multi Modal Balance Training Only
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 6/9 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi Modal Balance Training & Weight Loss (N=9) | Multi Modal Balance Training Only (N=11)
Fall (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (6)
Carpal Tunnel Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Car accident (General disorders) | 1 (1) | 0 (0)
Right knee swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Back/hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Hypoglycemia (Hepatobiliary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Conduct of the study was severely impacted by Coronavirus disease (COVID-19) as this study involved center-based exercise. All of the study participants stopped exercising and we were unable to obtain post-intervention outcome data for the longer time points that were proposed in the grant and even the short term outcome data was severely limited and underpowered. Due to their functional limitations the interventions were more labor intensive than had been anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT02806336/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT02806336/ICF_001.pdf